CLINICAL TRIAL: NCT07213544
Title: Comparison of Remimazolam Versus Propofol for Monitored Anesthetic Care in Elective Fractional Ablative CO₂ Laser
Brief Title: Remimazolam vs Propofol in Laser Burn Cases
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Principal Investigator, Rishi Patel, Assistant Professor-Faculty, Medical University of South Carolina
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: Pro00146765
Record Dates: First submitted 2025-09-22; First posted 2025-10-09 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Burn Scar; Hypertrophic Scarring; Procedural Sedation
MeSH Terms: conditions — Cicatrix, Hypertrophic | interventions — Propofol

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Remimazolam followed by Propofol (Active Comparator): Patients will be randomized to receive Remimazolam 0.075 mg/kg (maximum of 5 mg) for sedation during their first laser therapy session, then 4-6 weeks later at their next laser therapy session they will receive propofol 0.8 mg/kg IV bolus for sedation.
  Interventions: Drug: Remimazolam besylate; Drug: Propofol
- Propofol followed by Remimazolam (Active Comparator): Patients will be randomized to receive Propofol 0.8 mg/kg IV bolus for sedation during their first laser therapy session, then 4-6 weeks later at their next laser therapy session they will receive Remimazolam 0.075 mg/kg (maximum of 5 mg) for sedation.
  Interventions: Drug: Remimazolam besylate; Drug: Propofol

INTERVENTIONS:
Drug: Remimazolam besylate — Remimazolam
Drug: Propofol — Propofol

SUMMARY:
This randomized, single-blind, crossover study compares remimazolam and propofol for monitored anesthetic care during fractional ablative CO₂ laser therapy for burn scars. The primary aim is to assess incidence of respiratory depression, defined as a need for advanced airway maneuvers (jaw thrust/chin lift, insertion of oral or nasal airway, or bag mask ventilation), and hypopnea (respiratory rate < 8).

DETAILED DESCRIPTION:
Patients will be randomized to receive either remimazolam or propofol during their first laser session, and the alternate drug during their second session 4-6 weeks later. Outcomes include respiratory depression, sedation onset and recovery times, hemodynamic changes, and patient satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Undergoing both outpatient Session #1 and Session #2 of fractional ablative CO2 laser therapy

Exclusion Criteria:

* History of previous fractional ablative laser therapy for burn scar
* Procedure expected to last longer than 30 minutes
* Allergy such as dextran 40 or contraindication to either of the study drugs
* Pregnant and/or breastfeeding
* Subjects who are unable to or choose not to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Estimated)
Dates: Start 2025-11-12 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of respiratory depression | up to 24 hours after procedure ends
  The incidence of respiratory depression will include need for advanced airway maneuvers, or hypopnea events. Advanced airway maneuvers during the laser therapy procedure may include jaw thrust, chin lift, insertion of oral or nasal airway, or bag mask ventilation. A hypopnea event is defined as a respiratory rate <8.

SECONDARY OUTCOMES:
Time from initiation of sedation to peak sedation | up to 24 hours after procedure ends
  Time from initiation of sedation to peak sedation will be measured in minutes and calculated from the start time of induction to peak sedation when patient reaches a Modified Observer's Assessment of Alertness/Sedation (MOAA/S) score of less than 3. The MOAA/S scale ranges from 0 to 5, with higher scores indicating greater alertness and lower scores indicating deeper sedation:
  5: Responds readily to name spoken in a normal tone. 4: Lethargic response to name spoken in a normal tone. 3: Responds only after name is called loudly or repeatedly. 2: Responds only after mild prodding or shaking.
  1: Responds only after a painful trapezius squeeze. 0: Does not respond to a painful trapezius squeeze.
Time of cessation of sedation to full recovery | up to 24 hours after procedure ends
  Time of cessation of sedation to full recovery will be evaluated in minutes by marking when the last dose of anesthetic medication is given (cessation of sedation), to when the patient has reached full recovery from anesthesia. Full recovery from anesthesia is defined as when the patient reaches a Modified Observer's Assessment of Alertness/Sedation (MOAA/S) score ≥ 4.
  The MOAA/S scale ranges from 0 to 5, with higher scores indicating greater alertness and lower scores indicating deeper sedation:
  5: Responds readily to name spoken in a normal tone. 4: Lethargic response to name spoken in a normal tone. 3: Responds only after name is called loudly or repeatedly. 2: Responds only after mild prodding or shaking.
  1: Responds only after a painful trapezius squeeze. 0: Does not respond to a painful trapezius squeeze.
Cessation of sedation to full recovery | up to 24 hours after the procedure ends
  Cessation of sedation to full recovery will also be evaluated as length of PACU stay. This will be measured from the time the patient left the procedure room, to the time they are ready for discharge (marked as procedural care complete).
Satisfaction with Anesthesia | up to 24 hours after the procedure ends
  Satisfaction with Anesthesia will be measured using the Iowa Satisfaction with Anesthesia Scale (ISAS) approximately 15 minutes to two hours after arrival to to the recovery unit. This measures their satisfaction with Monitored Anesthesia Care (MAC).
  ISAS is an 11-item questionnaire designed to measure the satisfaction with monitored anesthesia care. The ISAS score is the mean of responses to all 11 questions. The score ranges from a minimum of -3 to a maximum of +3 when averaged together. The responses are: -3 = disagree very much, -2 = disagree moderately, -1 = disagree slightly, 1 = agree slightly, 2 = agree moderately, and 3 = agree very much. A score of +3 would imply a completely satisfied patient.
Felling pain on injection of sedation medication | up to 24 hours after the procedure ends
  Subjects will be asked if they felt pain upon the injection of the sedation medications, and will answer "yes" or "no". This will be asked at least 15 minutes after arriving to the recovery area after the procedure. "No" indicates they did not feel pain upon injection which means a better outcome.

OTHER OUTCOMES:
Incidence of hypotension | up to 24 hours after the procedure ends
  Incidence of hypotension during the procedure will measured by the use of vasopressors such as Norepinephrine or equivalent, as well as the lowest blood pressure reading during the procedure.
Incidence of low EtCO2 | up to 24 hours after the procedure ends
  Incidence of low EtCO2 will be measured by recording the lowest intraoperative EtCO2 reading during the procedure.
Incidence of hypoxemia | up to 24 hours after the procedure ends
  Baseline SpO2 and lowest SpO2 will be recorded to evaluate incidence of hypoxemia during the procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Rishi Patel, MD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No